CLINICAL TRIAL: NCT01182870
Title: Vitamin D and the Influenza Epidemic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Rolf Jorde, University of Tromsø
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UIT-ENDO-2010-1
Record Dates: First submitted 2010-08-11; First posted 2010-08-17 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: vitamin D; influenza; prevention
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cholecalciferol (Experimental): cholecalciferol in doses 800-6000 IU per day
  Interventions: Drug: choleclaciferol
- placebo (Placebo Comparator): placebo identical looking as cholecalciferol capsules
  Interventions: Drug: choleclaciferol

INTERVENTIONS:
Drug: choleclaciferol — 800-6000 IU cholecalciferol per day

SUMMARY:
Subjects included in ongoing vitamin d intervention trials were asked by questionnaire if they were ill with influenza during the winter season 2009/2010 to see if vitamin d supplementation prevented flu like disease.

ELIGIBILITY:
Inclusion Criteria:

* participant in vitamin D versus placebo study

Exclusion Criteria:

* none

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
influenza during the winter season 2009/2010 | up to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: rolf Jorde, md, Principal Investigator — University of Tromso, Norway
Locations (1):
- University of Tromsø, Tromsø, Tromsø, Norway